CLINICAL TRIAL: NCT04768699
Title: A Dose-ascending Study to Evaluate the Pharmacokinetics and Pharmacodynamics (PK/PD) of Recombinant Human Coagulation Factor VIIa for Injection in Patients With Hemophilia.
Brief Title: Study of Recombinant Human Coagulation Factor VIIa for Injection (FⅦa) in Patients With Hemophilia.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TQG203-I-01
Record Dates: First submitted 2021-01-29; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor
MeSH Terms: interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQG203(30µg/kg) (Experimental)
  Interventions: Drug: TQG203
- TQG203(90µg/kg) (Experimental)
  Interventions: Drug: TQG203/NovoSeven®
- NovoSeven®(90µg/kg) (Active Comparator): NovoSeven®,manufactured by Novo Nordisk Inc.
  Interventions: Drug: TQG203/NovoSeven®
- TQG203(180µg/kg) (Experimental)
  Interventions: Drug: TQG203

INTERVENTIONS:
Drug: TQG203 — TQG203,30µg/kg body weight, will be administered as intravenous (i.v.) administration over a period about 2minutes (min) on Study Day 1 once.
  Arms: TQG203(30µg/kg)
Drug: TQG203/NovoSeven® — In each of the two study periods (separated by a washout about two days),a single dose of TQG203 or NovoSeven® will be administered.TQG203 or NovoSeven®,90µg/kg body weight, will be administered as intravenous (i.v.) administration over a period about 2minutes (min) on Study Day 1.
  Arms: NovoSeven®(90µg/kg); TQG203(90µg/kg)
Drug: TQG203 — TQG203,180µg/kg body weight, will be administered as intravenous (i.v.) administration over a period about 2minutes (min) on Study Day 1 once.
  Arms: TQG203(180µg/kg)

SUMMARY:
Aim of this trial is to assess the pharmacokinetics and pharmacodynamics (PK/PD) of recombinant human coagulation factor VIIa for injection (FⅦa) in patients with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as congenital hemophilia A or B, and meet the following conditions: a. FⅧ<1% or FIX activity<2%; b. FⅧ inhibitor or FⅨ inhibitor titer in the screening period>5 BU (Nijmegen modified Bethesda method of detection).
* Age ≥18 and ≤75 years, male or female.
* No other drugs for the treatment of hemophilia have been used within 48 hours (2 days) before administration, including prothrombin complex and any FVII products, cryoprecipitate, fresh plasma and whole blood, etc.
* No obvious bleeding symptoms during PK medication (no active bleeding).
* Subjects of childbearing age agree to take effective contraceptive measures throughout the trial period, and continue to 28 days after the last medication.
* Volunteer to participate in this study, sign an informed consent form, have good compliance, and be able to cooperate with the experimental observation.

Exclusion Criteria:

* Any other bleeding disease except Congenital hemophilia A or B.
* Patients with any previous medical history or symptoms of arterial or venous thromboembolic events (such as atherosclerosis, myocardial infarction, ischemic stroke, transient ischemic attack, deep vein thrombosis or pulmonary hypertension embolism) or disseminated intravascular coagulation (DIC).
* Baseline and previous values of FⅦ inhibitor or rFVIIa inhibitor is positive.
* Vitamin K deficiency.
* Human immunodeficiency virus (HIV) positive and cluster of differentiation 4 (CD4) count ≤200/μl, the number of virus carriers ≥200 particles/μl or ≥400000 copies/ml.
* Subjects plan to perform elective surgery during the trial period.
* Those who are allergic to test drugs or any excipients.
* Severe anemia and need blood transfusion.
* Platelet count <80×10^9/L.
* Obvious liver or kidney damage: ALT or AST>2.5×ULN, or total bilirubin>1.5×ULN or serum creatinine>1.5×ULN.
* Have a history of cardiac surgery and need anticoagulation therapy; severe heart disease, including myocardial infarction, cardiac insufficiency grade 3 or above, the current New York Heart Association cardiac function grade II-IV.
* Hypertension that cannot be controlled with drug treatment: systolic blood pressure> 150 mmHg or diastolic blood pressure> 90 mmHg.
* Participated in other clinical studies (except FVIIa, FⅧ and FⅨ trials) within one month before the first medication.
* Diagnosed with hereditary diseases such as fructose intolerance, glucose malabsorption or sucrose-maltase deficiency.
* Alcoholism, drug abuse, mental disorders, other severe acute or chronic diseases, greater abnormal laboratory values, and those who are considered unsuitable by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic assessment, based on plasma concentration of Recombinant Human Coagulation Factor VIIa. | pre-dosing on Day 1 up to 24 hours post-dosing
Pharmacodynamic assessment, based on changes of activated partial thromboplastin time (APTT). | pre-dosing on Day 1 up to 24 hours post-dosing
Pharmacodynamic assessment, based on changes of prothrombin time (PT). | pre-dosing on Day 1 up to 24 hours post-dosing

SECONDARY OUTCOMES:
Immunogenicity assessment, based on inhibitors to Factor VIIa (FVIIa) or Factor VIII (FVIII) or Factor IX (FIX). | through study completion,an average of 1year.
Adverse events | The presence of adverse events will be observed, reported and sufficiently handled during subjects' participation in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China